CLINICAL TRIAL: NCT02510352
Title: Cohort of Patients With a Symptomatic Rotator Cuff Tear Treated Without Surgical Repair
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 0501079; DGOS (Other: 2006/040)
Record Dates: First submitted 2015-07-24; First posted 2015-07-29 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator cuff tear; MRI
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Rotator cuff tear: patients with a symptomatic rotator cuff tear treated without surgical repair

SUMMARY:
In accordance with national guidelines surgical repair of rotator cuff tear is the first-line strategy only in young patients, depending on tear size, fatty infiltration of rotator cuff muscles and articular status. In appropriate situations, a satisfactory result is expected in more than 80% of cases with a very good long-term outcome. On the other hand, the first-line strategy in older patients is conservative as the main objective is the treatment of pain and stiffness of the shoulder which can be achieved at least in the short-term with general and local medications and physiotherapy. In addition, poor prognostic factors such as massive tears and muscle fatty infiltration or atrophy, are more frequently present in those patients, leading to poor results of surgical treatment and a high risk of iterative tear after repair.

Because of a lack of evaluation, there is currently no identified prognostic factor of medical treatment and on the other hand no clinical situation in which a surgical repair is mandatory. Therefore, investigator designed this study as an observatory with the follow up of patients with a symptomatic rotator cuff tear treated conservatively.

DETAILED DESCRIPTION:
Patients are regularly monitored in rheumatology consultation at 3 months, 6 months, 1 year, 2 years, 30 months, 3 Years, 42 months, 4 years, 54 months and 5 years supplemented by simple radiological monitoring and an MRI followed by 1 year, 2 years and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Having a clinical symptoms suggesting a rotator cuff tear.
* Having a full-thickness tear of the rotator cuff confirmed by MRI.
* Covered by the Social Security system.

Exclusion Criteria:

* Being included in another clinical trial with a potential alteration of shoulder pathology management.
* Having a partial tear of the rotator cuff.
* Having a single lesion of the bicipital tendon.
* Having a traumatic tear of the rotator cuff less than 3-month old.
* Having surgery for rotator cuff tear planned within 3 months.
* Unable to understand the study protocol.
* Having a contra-indication to MRI.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having a full-thickness tear of the rotator cuff confirmed by MRI
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2006-04; Primary Completion 2009-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Functional evolution of patients with a rotator cuff tear | at 5 years
  Score to the Algo functional Constant score

SECONDARY OUTCOMES:
Assessing the radiological evolution of tenomuscular lesions induced by a rotator cuff tear | at 2 years
  lesion size measured by RMI
Assessing the radiological evolution of tenomuscular lesions induced by a rotator cuff tear | at 5 years
  lesion size measured by RMI
Functional evolution of patients with a rotator cuff tear | at 2 years
  Score to the Algo functional Constant score

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Thomas, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (12):
- France (12):
  - Hopital Ambroise Pare, Boulogne-Billancourt
  - Centre de Rhumatologie, Grenoble
  - Clinique Orthocèdres, Grenoble
  - Hopital Corentin-Celton, Issy-les-Moulineaux
  - Clinique Du Parc, Lyon
  - Centre Orthopedique Santy, Lyon
  - Cabinet de Rhumatologie, Marseille
  - Hopital Lariboisiere, Paris
  - Hopital Cochin, Paris
  - Chu de Saint Etienne, Saint-Etienne
  - Chu de Strasbourg, Strasbourg
  - Chu de Tours, Tours